CLINICAL TRIAL: NCT00446238
Title: Treatment of Depressed Adolescents With Physical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Harvard University (Other); Boston Children's Hospital (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Eva Szigethy, Associate Professor of Psychiatry, Pediatrics, and Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1K23MH064604-01A1 (NIH)
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Inflammatory Bowel Disease; Depression
Keywords: Depression; Physical Illness; Inflammatory Bowel Disease; Cognitive Behavioral Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): CBT enhanced with physical illness narrative, family education, and social skills components.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Standard of Community Care Treatment (Active Comparator): Standard of Community Care Treatment
  Interventions: Behavioral: Standard of Community Care Treatment

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — CBT enhanced with physical illness narrative, family education, and social skills components.
  Arms: Cognitive Behavioral Therapy
Behavioral: Standard of Community Care Treatment — Treatment as usual for depression and related symptoms provided within the community.
  Arms: Standard of Community Care Treatment

SUMMARY:
The purpose of this study is a randomized trial of cognitive-behavioral intervention (CBI) for eligible adolescents who have Inflammatory Bowel Disease and subsyndromal depressive symptoms, but who did not meet diagnostic criteria for major depressive disorder at the time of randomization into the study.

Hypotheses

1. This preliminary randomized trial will demonstrate the feasibility of a large-scale research initiative.
2. Subjects will experience no adverse events, and the CBI group will demonstrate improved negative cognitions, depressive symptomatology, and functioning at the post-intervention and 6- through 12-month follow-ups.

DETAILED DESCRIPTION:
This study is a pilot study, which will serve to determine the feasibility of a larger research initiative. The broader research is aimed at the prevention of depressive disorders in adolescents with inflammatory bowel disease (IBD) who have risk factors for depression, using a psychotherapeutic intervention. The intervention is based on a cognitive-behavioral approach to treating depression, the Primary and Secondary Control Enhancement Training (PASCET), that has been modified and enhanced with physical illness narrative, social skills, and family components (PASCET-Physical Illness), to make it more appropriate for physically ill adolescents at risk for major depression. The cognitive-behavioral intervention (CBI) draws on an etiological hypothesis that depression in adolescents with chronic physical illness results from cumulative risk factors such as distorted cognitive processes, negative physical illness experience, poor social functioning, and ineffective family interactions. Thus, the development of depression may be prevented by teaching adolescents effective strategies to 1) cope using cognitive-behavioral skills, 2) enhance social functioning, 3) develop a more cohesive illness narrative, and 4) improve family communication skills.

The study is a randomized trial of the CBI for adolescents with IBD and depressive symptoms, using the provision of psychoeducational materials as the attention control group. This study is a pilot study designed to show feasibility of assessing and treating youth with sub-syndromal depressive symptoms and IBD using a randomized clinical design at Children's Hospital Pittsburgh (CHP) as a preliminary step for designing a two-site randomized trial Children's Hospital of Pittsburgh and Children's Hospital Boston powered to test preventive effects of this CBI in this medically co-morbid population.

In this study, eligible adolescents who are at risk for developing depression due to having a chronic physical illness (IBD) as well as having subsyndromal depressive symptoms but who do not currently meet diagnostic criteria for major depressive disorder according to a diagnostic interview will be randomly assigned either to receive CBI or psychoeducation.

ELIGIBILITY:
Inclusion Criteria:

* Step One

  1. Ages 11 to 17 inclusive.
  2. Capable of completing CDI
  3. English-speaking.
  4. Meeting diagnostic criteria for IBD (The date of diagnosis = date of the first diagnostic test confirming IBD)
  5. Absence of mental retardation by history
  6. Having at least one appointment at the gastroenterology clinic at CHP.
* Step Two: Assessment

  1) CDI and/or CDI-P equal to or more than 9 at Step 1
* At Intervention Phase

  1. CDI score equal to or more than 9 AND/OR CDI-P score equal to or more than 9 at T0.
  2. Absence of recent suicide attempt (within one month of study enrollment) or depression severity requiring acute psychiatric hospitalization),
  3. Age 11-17 years inclusive,
  4. Presence of at least one biological parent.

Exclusion Criteria:

1. Current major depression or dysthymia by Diagnostic and Statistical Manual (DSM)-IV criteria
2. History or current episode of bipolar disorder, eating disorder, or psychotic disorder by DSM-IV criteria.
3. Mental retardation by history
4. Antidepressant or stimulant medications within one month of assessment
5. Suicidality with plan or of severity requiring immediate psychiatric hospitalization or significant act involving intentional self-harm, e.g. cutting or overdose, resulting in medical attention.
6. Unacceptable risk for dangerousness to others as indicated by homicidal (or other violent) ideation, intent or plan or action, or use of illegal weapons.
7. Current pregnancy by history.
8. Substance abuse within one month of enrollment other than nicotine dependence.
9. Current treatment with cognitive behavioral therapy (CBT) or failure of previous CBT trial for depression judged adequate by at least 12 treatment sessions over a period of less than 1 year conducted by an appropriately trained mental health provider.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2002-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in CDI at 14 weeks | Week 0, Week 14
  Change in Childhood Depression Inventory (CDI) scores from week 0 to study endpoint, week 14

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szigethy, MD, PhD, Principal Investigator — University of Pittsburgh / Children's Hospital of Pittsburgh; David DeMaso, MD, Principal Investigator — Harvard University / Children's Hospital Boston
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Szigethy E, Carpenter J, Baum E, Kenney E, Baptista-Neto L, Beardslee WR, Demaso DR. Case study: longitudinal treatment of adolescents with depression and inflammatory bowel disease. J Am Acad Child Adolesc Psychiatry. 2006 Apr;45(4):396-400. doi: 10.1097/01.chi.0000198591.45949.a4. PMID 16601643
- [Result] Szigethy E, Whitton SW, Levy-Warren A, DeMaso DR, Weisz J, Beardslee WR. Cognitive-behavioral therapy for depression in adolescents with inflammatory bowel disease: a pilot study. J Am Acad Child Adolesc Psychiatry. 2004 Dec;43(12):1469-77. doi: 10.1097/01.chi.0000142284.10574.1f. PMID 15564816
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Szigethy E, Kenney E, Carpenter J, Hardy DM, Fairclough D, Bousvaros A, Keljo D, Weisz J, Beardslee WR, Noll R, DeMASO DR. Cognitive-behavioral therapy for adolescents with inflammatory bowel disease and subsyndromal depression. J Am Acad Child Adolesc Psychiatry. 2007 Oct;46(10):1290-1298. doi: 10.1097/chi.0b013e3180f6341f. PMID 17885570